CLINICAL TRIAL: NCT07333118
Title: A Clinical Study to Evaluate the Safety and Efficacy of GT801 Injection in the Treatment of Moderate-to-Severe Refractory Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-801-002
Record Dates: First submitted 2025-12-15; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Moderate to Severe Refractory Autoimmune Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT801 Injection treatment group (Experimental): GT801 Injection
  Interventions: Biological: GT801 Injection

INTERVENTIONS:
Biological: GT801 Injection — GT801 Injection

SUMMARY:
This is a single-arm, open-label, dose-escalation and dose-expansion clinical trial designed to evaluate the safety, efficacy, and cellular metabolism kinetics of GT801 in the treatment of moderate-to-severe refractory autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* 1. The participant or their legal representative voluntarily signs a written informed consent form and is willing and able to comply with the study procedures.
* 2. Aged 18 to 65 years old (inclusive) at the time of signing the informed consent, regardless of gender.
* 3. Participants with Systemic Lupus Erythematosus (SLE) must meet the following criteria:
* a) Fulfill the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria for SLE.
* b) Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2000) score ≥ 6, with at least one British Isles Lupus Assessment Group Index (BILAG-2004) Grade A (severe manifestation) or two Grade B (moderate manifestation) organ scores, or both; or SLEDAI-2000 score ≥ 8.
* c) Meet the definition of refractory or relapsing disease: No response to conventional treatment for more than 6 months, or disease reactivation after achieving remission. Conventional treatment is defined as the use of glucocorticoids and cyclophosphamide plus at least one of the following immunomodulatory agents: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents including rituximab, belimumab, and tabalumab.
* 4. Participants with Idiopathic Inflammatory Myopathy (IIM) must meet the following criteria:
* a) Fulfill the 2017 EULAR/ACR classification criteria for inflammatory myopathy (including Dermatomyositis [DM], Polymyositis [PM], Antisynthetase Syndrome [ASS], and Necrotizing Myopathy [NM]).
* b) Positive for myositis-specific antibodies or myositis-associated antibodies.
* c) Must have moderate to severe IIM at screening, defined as Manual Muscle Testing-8 (MMT-8) score ≥ 142, or MMT-8 score < 142 plus meeting 2 of the following criteria:
* 1) Physician Global Assessment (PGA) (Visual Analog Scale [VAS]) ≥ 2 cm (on a 10-cm VAS).
* 2) Patient Global Assessment (PtGA) (VAS) ≥ 2 cm (on a 10-cm VAS).
* 3) Health Assessment Questionnaire (HAQ) score > 0.25.
* 4) Elevation of one or more muscle enzymes (creatine kinase [CK], lactate dehydrogenase [LDH], aspartate aminotransferase [AST], alanine aminotransferase [ALT]) ≥ 1.5 × Upper Limit of Normal (ULN).
* d) Meet the definition of refractory/relapsing or progressive disease:
* 1) Refractory/relapsing: No response to conventional treatment for more than 6 months, or disease reactivation after achieving remission. Conventional treatment is defined as the use of glucocorticoids and cyclophosphamide plus at least one of the following immunomodulatory agents: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents including rituximab, belimumab, and tabalumab.
* 2) Progressive: Development of worsening myositis or rapidly progressive interstitial lung disease.
* 5. Participants with Systemic Sclerosis (SSc) must meet the following criteria:
* a). Fulfill the 2013 American College of Rheumatology (ACR) classification criteria for SSc.
* b). Positive for SSc-related autoantibodies.
* c). Meet the definition of refractory/relapsing or progressive disease:
* 1) Refractory/relapsing: No response to conventional treatment for more than 6 months, or disease reactivation after achieving remission. Conventional treatment is defined as the use of glucocorticoids and cyclophosphamide plus at least one of the following immunomodulatory agents: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents including rituximab, belimumab, and tabalumab.
* 2) Refractory/relapsing: No response to conventional treatment for more than 6 months, or disease reactivation after achieving remission. Conventional treatment is defined as the use of glucocorticoids and cyclophosphamide plus at least one of the following immunomodulatory agents: antimalarials, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents including rituximab, belimumab, and tabalumab.
* 6. Participants with ANCA-Associated Vasculitis (AAV) must meet the following criteria:
* a). Fulfill the 2022 ACR/EULAR classification criteria for ANCA-associated vasculitis, including Microscopic Polyangiitis (MPA), Granulomatosis with Polyangiitis (GPA), and Eosinophilic Granulomatosis with Polyangiitis (EGPA).
* b). Positive for ANCA-related antibodies (myeloperoxidase-ANCA [MPO-ANCA] or proteinase 3-ANCA [PR3-ANCA]).
* c). Birmingham Vasculitis Activity Score (BVAS) ≥ 15 points (total score: 63 points), indicating active vasculitis.
* d). Meet the definition of refractory/relapsing disease: No response to conventional treatment for more than 6 months, or disease reactivation after achieving remission. Conventional treatment is defined as the use of glucocorticoids and cyclophosphamide plus at least one of the following immunomodulatory agents: antimalarials, azathioprine, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents including rituximab, belimumab, and tabalumab.
* 7. Participants with Sjogren's Syndrome must meet the following criteria:
* a). Fulfill the 2002 American-European Consensus Group (AECG) criteria for primary Sjogren's Syndrome or the 2016 ACR/EULAR classification criteria.
* b). EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) score ≥ 6.
* c). Positive for anti-SSA/Ro antibodies.
* d). Meet the definition of refractory/relapsing disease: No response to conventional treatment for more than 6 months, or disease reactivation after achieving remission. Conventional treatment is defined as the use of glucocorticoids and cyclophosphamide plus at least one of the following immunomodulatory agents: antimalarials, azathioprine, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents including rituximab, belimumab, and tabalumab.
* 8. Laboratory test results at screening must meet the following criteria (excluding indicators related to the study disease):
* a). Absolute neutrophil count ≥ 1.5 × 10⁹/L.
* b). Hemoglobin ≥ 80 g/L; Platelet count ≥ 50 × 10⁹/L.
* c). Alanine Aminotransferase (ALT) ≤ 3 × ULN; Aspartate Aminotransferase (AST) ≤ 3 × ULN (unless elevations of ALT and/or AST are assessed by the investigator to be related to Polymyositis [PM] or Dermatomyositis [DM]); Total Bilirubin (TBIL) < 2 × ULN (for participants with Gilbert's syndrome, Direct Bilirubin [DBIL] ≤ 1.5 × ULN).
* d). Creatinine clearance rate ≥ 30 mL/min.
* e). Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN; Prothrombin Time (PT) ≤ 1.5 × ULN.
* f). Left Ventricular Ejection Fraction (LVEF) ≥ 50% confirmed by echocardiography, with no clinically significant electrocardiogram (ECG) abnormalities detected.
* g). Baseline oxygen saturation > 92% measured on room air.
* 9. Women of childbearing potential must:
* a). Have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result at screening, confirmed by the investigator.
* b). Agree to avoid breastfeeding during study participation until at least 1 year after GT801 injection or until GT801 cells are no longer detectable by two consecutive flow cytometry tests, whichever is later.
* c). Male participants with sexual partners and female participants of childbearing potential must agree to use highly effective contraceptive methods (e.g., oral contraceptives, intrauterine devices, or condoms) starting from screening until at least 1 year after GT801 injection or until GT801 cells are no longer detectable by two consecutive flow cytometry tests, whichever is later. Male participants must agree to use condoms during sexual contact with pregnant women or women of childbearing potential for at least 1 year after GT801 injection, even after successful vasectomy.

Exclusion Criteria:

* 1. Participants with SLE
* a. Drug-induced systemic lupus erythematosus.
* b. Participants with lupus crisis; or those with concurrent diseases requiring the use of protocol-prohibited drugs, who are deemed ineligible for enrollment by the investigator.
* 2. Participants with IIM
* a. Documented inclusion body myositis (IBM), drug-induced polymyositis (PM) or dermatomyositis (DM), malignancy-associated PM or DM, or non-inflammatory myopathies (e.g., muscular dystrophy).
* b. Uncontrolled extramuscular disease manifestations related to PM or DM:
* 1) ILD: Forced vital capacity (FVC) < 55% or requirement for oxygen therapy.
* 2) Severe dysphagia manifestations that, in the investigator's judgment, would increase the participant's risk of participating in the clinical trial.
* 3) Severe cardiac manifestations (e.g., congestive heart failure, cardiac arrhythmia, conduction abnormalities requiring treatment, or myocardial infarction) that, in the investigator's judgment, would increase the participant's risk of participating in the clinical trial.
* 3. Participants with SSc
* a. Severe SSc-associated pulmonary arterial hypertension (PAH) that is uncontrollable with medical treatment.
* b. Rapidly progressive SSc-related lower gastrointestinal tract (small and large intestine) involvement requiring parenteral nutrition; active gastric antral vascular ectasia.
* c. Uncontrolled or rapidly progressive ILD with oxygen saturation (SaO₂) < 92% (on room air at rest); or requirement for mechanical ventilation support within 1 year prior to signing the informed consent form.
* 4. Participants with ANCA-Associated Vasculitis (AAV)
* a. Presence of rapidly progressive glomerulonephritis, acute mononeuritis multiplex, or central nervous system (CNS) involvement unrelated to AAV at screening.
* b. Life-threatening severe vasculitis (including diffuse alveolar hemorrhage, respiratory failure, intestinal perforation or massive hemorrhage, cerebral vasculitis, cardiac vasculitis, etc.).
* c. Secondary vasculitis (e.g., systemic lupus erythematosus, Henoch-Schönlein purpura, drug-induced, malignancy-related, infection-related, primary immunodeficiency, etc.).
* 5. Participants with Sjögren's Syndrome (SS)
* a. Presence of poorly controlled severe systemic primary Sjögren's disease (pSjD) manifestations at baseline that, in the investigator's assessment, would place the participant at excessive risk, including pSjD-associated cytopenia of Grade ≥ 2 per the Common Terminology Criteria for Adverse Events (CTCAE).
* b. Secondary Sjögren's syndrome with a primary diagnosis of other confirmed autoimmune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, scleroderma, and inflammatory bowel disease).
* c. Regular use of medications known to cause xerostomia/keratoconjunctivitis sicca (a common major side effect).
* d. Concomitant diseases that may interfere with the efficacy assessment of primary Sjögren's syndrome, e.g., inflammatory bowel disease, gout, sarcoidosis, amyloidosis, graft-versus-host disease, IgG4-related disease, etc.

All Participants:

* 6. History of severe hypersensitivity reactions or allergies.
* 7. Detection of pre-existing anti-polyethylene glycol (anti-PEG) antibodies in the body prior to GT801 infusion.
* 8. Contraindications to or hypersensitivity reactions to any component of the investigational product.
* 9. History of the following cardiac diseases:
* a. New York Heart Association (NYHA) Class III or IV congestive heart failure.
* b. Myocardial infarction or coronary artery bypass grafting within 6 months prior to screening.
* c. History of clinically significant ventricular arrhythmia or unexplained syncope not caused by vasovagal response or dehydration; or corrected QT interval (QTc) > 480 ms at screening; history of severe non-ischemic cardiomyopathy.
* 10. History of any active malignancy or malignant tumor within 5 years prior to screening, except for the following conditions: early-stage tumors treated with curative intent (carcinoma in situ or Stage I tumors, non-ulcerative primary melanoma with depth < 1 mm and no lymph node involvement), basal cell carcinoma of the skin, squamous cell carcinoma of the skin, cervical carcinoma in situ, or ductal carcinoma in situ of the breast that has undergone potentially curative treatment.
* 11. Any other known autoimmune diseases besides the study disease.
* 12. Long-term use of anticoagulant drugs that affect coagulation function.
* 13. Clinically significant bleeding symptoms or confirmed bleeding tendency within 6 months prior to screening (e.g., gastrointestinal bleeding, hemorrhagic gastric ulcer, etc.); hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophilia, coagulation disorders, hypersplenism, etc.); arterial or venous thrombotic events within 6 months prior to screening (e.g., cerebrovascular diseases including cerebral hemorrhage and cerebral infarction, deep vein thrombosis, and/or pulmonary embolism).
* 14. Presence of severe underlying medical conditions at screening, such as:
* a. Evidence of uncontrolled viral, bacterial, fungal, or other infections requiring systemic intravenous therapy.
* b. Clear clinical evidence of dementia or altered mental status.
* c. History of any other central nervous system diseases or neurodegenerative disorders (e.g., epilepsy, convulsions, paralysis, aphasia, stroke, severe traumatic brain injury, dementia, Parkinson's disease, psychosis).
* 15. Positive results for any of the following tests:
* a. Human Immunodeficiency Virus (HIV) antibody positive.
* b. Hepatitis B surface antigen (HBsAg) positive; or hepatitis B core antibody (HBcAb) positive with hepatitis B virus (HBV)-DNA levels above the lower limit of quantification of the assay.
* c. Hepatitis C virus (HCV) antibody positive with HCV RNA levels above the lower limit of quantification of the assay.
* d. Syphilis antibody positive (excluding false-positive results caused by underlying diseases).
* 16. Positive results for cytomegalovirus (CMV) DNA or Epstein-Barr virus (EBV) DNA testing.
* 17. Active tuberculosis or latent tuberculosis that has not received appropriate treatment prior to screening.
* 18. Receipt of other investigational drugs within 4 weeks prior to signing the informed consent form (ICF); or the interval between the ICF signing date and the last dose of the previous clinical trial participation is still within 5 half-lives of the drug, whichever is longer.
* 19. Receipt of plasma exchange therapy or immunoadsorption therapy within 4 weeks prior to investigational product administration.
* 20. Receipt of B-cell-targeted drug therapy within 1 week prior to investigational product administration, including but not limited to rituximab, belimumab, tabalumab, etc.
* 21. Receipt of biologic therapy such as anti-TNF-α antibodies within 12 weeks prior to investigational product administration.
* 22. Use of tacrolimus, cyclosporine, azathioprine, mycophenolate mofetil, mycophenolic acid, methotrexate, etc., within 2 weeks prior to investigational product administration.
* 23. Receipt of neonatal Fc receptor (FcRn) antagonist therapy (e.g., efgartigimod, etc.) within 3 weeks prior to investigational product administration.
* 24. Receipt of complement inhibition therapy (e.g., eculizumab, etc.) within 3 weeks prior to investigational product administration.
* 25. Vaccination with live attenuated vaccines or mRNA vaccines within 8 weeks prior to enrollment; or inactivated vaccines within 4 weeks prior to enrollment.
* 26. Major surgery within 8 weeks prior to screening, or planned surgery during the study period.
* 27. History of organ transplantation.
* 28. Prior receipt of chimeric antigen receptor T-cell (CAR-T) therapy targeting any antigen.
* 29. Presence of any conditions that, in the investigator's judgment, would prevent the participant from completing the entire trial, confound trial results, or make trial participation not in the participant's best interest.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing dose limiting toxicity | 28 days
  The proportion of participants with dose-limiting toxicity (DLT) occurring within 28 days after infusion
Adverse Events (AEs) occurring after infusion and their proportions | 3 months
  Adverse Events (AEs) occurring after infusion and their proportions

SECONDARY OUTCOMES:
Efficacy outcomes for Systemic Lupus Erythematosus (SLE) | 1, 2, 3 and 6 Months post GT801 infusion
  SLE Response index 4(SRI-4) response: Min/Max Value: Not specified; a decrease in score indicates improvment, higher scores indicate worse outcome
Efficacy outcomes for Idiopathic Inflammatory Myopathies (IIM) | 1, 2, 3 and 6 Months post GT801 infusion
  Total lmprovement Score (TlS): Min/Max Value: Not specified; an increase in score indicates improvement, higher scores indicate better outcome.
Efficacy outcomes for Systemic Sclerosis (SSc) | 1, 2, 3 and 6 Months post GT801 infusion
  Combined Response Index in Systemic Sclerosis (CRISS): the score ranges from 0 to 1 point; a score ≥ 0.6 indicates treatment improvement, while a score < 0.6 indicates no disease improvement.
Efficacy Outcomes for ANCA-Associated Vasculitis (AAV) | 6 and 12 Months post GT801 infusion
  The proportion of subjects achieving complete remission and partial remission
Efficacy Outcomes for Participants with Sjogren's Syndrome | 6 and 12 Months post GT801 infusion
  ESSDAI response rates
Efficacy Outcomes for Participants with Sjogren's Syndrome | 6 and 12 Months post GT801 infusion
  ESSPRI response rates
Cellular Kinetics of All Participants: Time to Peak Expansion of GT801 Cells After Infusion (Tmax) | From infusion to 12 months
  Time to Peak Expansion (Tmax) refers to the time point at which the infused target cells proliferate to the peak quantity in the participants' bodies.
Cellular Kinetics of All Participants: Expansion Peak of GT801 Cells After Infusion (Cmax) | From infusion to 12 months
  Expansion Peak (Cmax) refers to the maximum quantity of infused GT801 cells achieved during their proliferation in the participants' bodies.
Cellular Kinetics of All Participants: Area Under the Curve (AUC) of GT801 Cells After Infusion | From infusion to 12 months
  Area Under the Curve (AUC) refers to the area enclosed by the curve of GT801 cell quantity change over time after infusion and the time axis.
Cellular Kinetics of All Participants: Duration of Detectable Concentration of GT801 Cells After Infusion (Tlast) | From infusion to 12 months
  Duration of Detectable Concentration (Tlast) refers to the time period from the infusion of GT801 cells to the last time point at which the target cells can be detected in the peripheral blood or target tissues.
Pharmacodynamic characteristics in participants for all participants | From infusion to 2 months
  Monitor serum cytokine levels after infusion

OTHER OUTCOMES:
Exploration of Peripheral Blood Lymphocyte Subsets and B Lymphocyte Subsets: Changes in T Cells and NK Cells | 1, 3, 6, 9 Months post GT801 infusion
  Determination of the counts of T cells and NK cells
Exploration of Peripheral Blood Lymphocyte Subsets and B Lymphocyte Subsets: Duration of B-Cell Depletion | 3, 6, 9 Months post GT801 infusion
  Determination of B-cell counts and calculation of the duration of B-cell count reduction
Exploration and analysis of BCR repertoire diversity via BCR sequencing | 1, 3, 6, 9 Months post GT801 infusion
  Detection of BCR diversity on B cells via sequencing
Pathological changes of involved organs before and after treatment | From GT801 infusion to 3 months
  Pathological examination of lesion tissue biopsies was performed to observe the changes in histopathological characteristics after treatment compared with those before treatment, such as fibrosis, vascular lesions, and inflammatory cell infiltration.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No